CLINICAL TRIAL: NCT05214066
Title: Prospective Study of Combined 4-Day ATG Regimen for Prophylaxis of aGVHD in Matched Sibling Donor PBSCT
Brief Title: Efficacy and Safety Study of 4-Day ATG Regimen for Prophylaxis of aGVHD in Matched Sibling Donor PBSCT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Daihong Liu, Director, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 81370667
Record Dates: First submitted 2022-01-17; First posted 2022-01-28 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-01

CONDITIONS: aGVHD; cGVHD
Keywords: ATG; Matched sibling donor; peripheral blood stem cell transplantation
MeSH Terms: interventions — thymoglobulin; Antilymphocyte Serum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 4-day ATG combined regimen (Experimental): ATG combined regimen for prophylaxis of GVHD, includes ATG, MMF (Mycophenolate mofetil), CsA (cyclosporin A) and MTX (methotrexate). All recipients in this arm received ATG, CsA, mycophenolate mofetil, and short-term methotrexate for GVHD prophylaxis. ATG (Thymoglobuline, rabbit) was used as 1 mg/kg/d from day -5 to day -3 and 2 mg/kg/d on day -2. CsA (3 mg/kg, q12h, i.v.) was used from day -9, and the concentration was adjusted to 180-200 ng/mL. CsA was switched to oral administration when the patient's bowel function recovered. From day -9, 0.5 g of mycophenolate mofetil was administered orally from every 12 h, which was withdrawn on day +30. After graft infusion, MTX was given for all patients at 15 mg/m2 on day +1 and 10 mg/m2 on days +3, +6 and +11.
  Interventions: Drug: Rabbit ATG

INTERVENTIONS:
Drug: Rabbit ATG — ATG (Thymoglobuline, rabbit) was used as 1 mg/kg/d from day -5 to day -3 and 2 mg/kg/d on day -2.
  Other Names: Thymoglobuline

SUMMARY:
The purpose of this study is to determine the efficacy and safety of combined ATG #antithymocyte globulin # regimen (5mg/kg divided from day -5 to day -2) for aGVHD(acute graft-versus-host disease ) prophylaxis in matched sibling donor peripheral blood stem cell transplantation (MSD-PBSCT).

DETAILED DESCRIPTION:
Transplantation with G-CSF #Granulocyte colony stimulating factor #mobilized peripheral blood stem cell (PBSCT) has been a stable transplant setting with matched sibling donor transplantation. Unmanipulated haploidentical donor PBSCT (haplo-PBSCT) has been applied in patients with hematologic malignancies. In our previous cohort study, haplo-PBSCT was associated with lower incidence of severe acute GVHD and extensive chronic GVHD compared with matched sibling donor PBSCT (MSD-PBSCT). Haplo-PBSCT has the same GVHD prophylaxis regimen with MSD-PBSCT, except ATG. It suggested the potential advantage of ATG in prophylaxis of GVHD and improvement of long term quality of life of the transplant recipients, which motivate us to observe the efficacy of combined ATG regimen for GVHD prophylaxis in MSD-PBSCT.

ELIGIBILITY:
Inclusion Criteria:

* Patients were aged from 14 to 65 years;
* Patients were diagnosed of acute leukemia or MDS;
* There were indications of MSD-PBSCT for these patients;
* Patients without any uncontrolled infections or without severe pulmonary, renal, hepatic or cardiac diseases.

Exclusion Criteria:

* Patients with any uncontrolled infections or with severe pulmonary,renal, hepatic or cardiac diseases;
* AML patients with t (15;17).

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with severe cGVHD | 1 year
  Chronic graft versus host disease grading criteria (refer to NIH criteria)

SECONDARY OUTCOMES:
Number of participants with aGVHD as assessed by acute graft versus host disease grading criteria (refer to Glucksberg criteria) | 100 days
  Cumulative incidence of aGVHD
OS | 1 year
  overall survival of enrolled patients
Number of participants relapse as assessed by NCCN (National Comprehensive Cancer Network )criteria | 1 year
  cumulative incidence of relapse
DFS | 1 year
  disease-free survival
NRM | 1 year
  non-relapse mortality

CONTACTS AND LOCATIONS:
Overall Officials: Daihong Liu, Doctor, Study Director — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China